CLINICAL TRIAL: NCT03158129
Title: Phase II Study of Induction Checkpoint Blockade for Untreated Stage I-IIIA Non-Small Cell Lung Cancers Amenable for Surgical Resection
Brief Title: Nivolumab With or Without Ipilimumab or Chemotherapy in Treating Patients With Previously Untreated Stage I-IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0982; NCI-2018-01210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0982 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stage I Lung Non-Small Cell Cancer AJCC v7; Stage IA Lung Non-Small Cell Carcinoma AJCC v7; Stage IB Lung Non-Small Cell Carcinoma AJCC v7; Stage II Lung Non-Small Cell Cancer AJCC v7; Stage IIA Lung Non-Small Cell Carcinoma AJCC v7; Stage IIB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Ipilimumab; CTLA-4 Antigen; Nivolumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (nivolumab) (Experimental): Participants receive nivolumab IV over 60 minutes on days 1, 15, and 29 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab
- Arm B (nivolumab, ipilimumab) (Experimental): Participants receive nivolumab as in Arm A and receive ipilimumab IV over 90 minutes on day 1 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab
- Arm C (nivolumab, cisplatin, docetaxel, pemetrexed) (Experimental): Patients receive nivolumab IV over 30 minutes and cisplatin IV over 2 hours on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel IV over 1 hour or pemetrexed IV over 10 minutes on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Biological: Nivolumab; Drug: Pemetrexed
- Arm D (ipilimumab, nivolumab, chemotherapy) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1, nivolumab IV over 30 minutes on days 1, 22, and 43, and cisplatin (or carboplatin) IV over 2 hours on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel IV over 1 hour or pemetrexed IV over 10 minutes on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Docetaxel; Biological: Ipilimumab; Biological: Nivolumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm D (ipilimumab, nivolumab, chemotherapy)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm C (nivolumab, cisplatin, docetaxel, pemetrexed); Arm D (ipilimumab, nivolumab, chemotherapy)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm C (nivolumab, cisplatin, docetaxel, pemetrexed); Arm D (ipilimumab, nivolumab, chemotherapy)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (nivolumab, ipilimumab); Arm D (ipilimumab, nivolumab, chemotherapy)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm C (nivolumab, cisplatin, docetaxel, pemetrexed); Arm D (ipilimumab, nivolumab, chemotherapy)

SUMMARY:
This phase II trial studies how well nivolumab works when given alone and in combination with ipilimumab or chemotherapy in treating patients with previously untreated stage I-IIIA non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cisplatin, docetaxel, and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab with ipilimumab or chemotherapy may work better in treating patients with non-small cell lung cancer compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the major pathologic response rate (MPRR) in patients treated with induction nivolumab, nivolumab plus ipilimumab, and nivolumab plus platinum-based chemotherapy.

SECONDARY OBJECTIVES:

I. Toxicity (assessed by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4).

II. Peri-operative morbidity and mortality. III. CD8 positive (+) tumor infiltrating lymphocytes (TILs) in resected tumor tissues of patients treated with nivolumab alone and nivolumab plus ipilimumab and nivolumab plus platinum-based chemotherapy.

IV. Quantification of CD8+ TILs will be assessed by counting the cells positive for staining with an anti-CD8 antibody by immunohistochemistry in five random square areas (1 mm^2 each) in both intratumoral and peritumoral compartments using the automated Aperio system.

V. Response rates to induction treatment (by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1).

VI. Recurrence-free survival. VII. Overall survival. VIII. To correlate major pathologic response with recurrence-free and overall survival.

IX. Complete resection (R0) rate. X. Pathologic complete response (pCR) in resected tumor specimens. XI. To correlate response assessed by imaging studies with outcomes (both major pathologic response to treatment and long-term recurrence-free survival).

XII. To correlate blood, tissue, and stool-based biomarkers with efficacy and toxicity.

EXPLORATORY OBJECTIVES:

I. To identify novel prognostic and predictive markers present at diagnosis. II. To determine modulation of markers by induction immunotherapy and/or immunotherapy plus platinum-based chemotherapy in order to inform future translational studies.

OUTLINE: Patients are randomized to Arms A and B and enrolled in Arm C or D after completion of enrollment to Arms A and B.

ARM A: Patients receive nivolumab intravenously (IV) over 60 minutes on days 1, 15, and 29 in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive nivolumab as in Arm A and receive ipilimumab IV over 90 minutes on day 1 in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive nivolumab IV over 30 minutes and cisplatin IV over 2 hours on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel IV over 1 hour or pemetrexed IV over 10 minutes on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive ipilimumab IV over 90 minutes on day 1, nivolumab IV over 30 minutes on days 1, 22, and 43, and cisplatin (or carboplatin) IV over 2 hours on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity. Patients also receive docetaxel IV over 1 hour or pemetrexed IV over 10 minutes on days 1, 22, and 43 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment and surgery, patients are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed previously untreated non-small cell lung cancer. If a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected lung cancer are eligible, but pathology must be confirmed prior to initiating treatment on study. Neuroendocrine carcinomas are not eligible. Carcinomas with neuroendocrine differentiation are eligible
* Patients with stage IA or stage IB < 4 cm (according to American Joint Committee on Cancer [AJCC] 7th edition) are eligible for randomization into arms A and B only. Patients with stage IB >= 4 cm, IIA, IIB, or IIIA disease (according to AJCC 7th edition) are eligible for randomization into arms A, and B, and for enrollment into arms C and D
* Patients with stage IIIA must not have more than one mediastinal lymph node station involved by tumor
* All patients must have lymph node evaluation of contralateral stations 2 and/or 4 to exclude N3 disease
* The patient must be a suitable candidate for surgery, in the opinion of the treating physician
* Signed and dated written informed consent must be provided by the patient prior to admission to the study in accordance with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines and to the local legislation
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 8.0 g/dL
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except subjects with Gilbert syndrome who can have total bilirubin < 3.0 mg/dL)
* Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 50 mL/min using Cockcroft-Gault formula for creatinine clearance calculation OR 24-hour urine creatinine clearance >= 50 mL/min

Exclusion Criteria:

* Prior systemic therapy or radiation therapy for treatment of the current lung cancer
* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug
* Pregnant or lactating female: Women of childbearing potential (WOCB) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of nivolumab; Women of childbearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* Unwillingness or inability to follow the procedures required in the protocol
* Patients with pre-existing sensorineural hearing impairment/loss or newly diagnosed as documented by an audiology assessment performed prior to study enrollment may not be eligible for cisplatin and may be dispositioned to carboplatin, as determined by the treating physician.
* Patients with a history of severe hypersensitivity reaction to taxotere and or polysorbate 80 must be excluded
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Prior treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody
* Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of severe hypersensitivity reaction to any monoclonal antibody and/or to study drug components
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Patients who are sexually active, with preserved reproductive capacity, and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during and after the trial
* Women of child bearing potential (WOCBP) should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug(s); Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; Women who are not of childbearing potential as well as azoospermic men do not require contraception
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cascone, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cascone T, Leung CH, Weissferdt A, Pataer A, Carter BW, Godoy MCB, Feldman H, William WN Jr, Xi Y, Basu S, Sun JJ, Yadav SS, Rojas Alvarez FR, Lee Y, Mishra AK, Chen L, Pradhan M, Guo H, Sinjab A, Zhou N, Negrao MV, Le X, Gay CM, Tsao AS, Byers LA, Altan M, Glisson BS, Fossella FV, Elamin YY, Blumenschein G Jr, Zhang J, Skoulidis F, Wu J, Mehran RJ, Rice DC, Walsh GL, Hofstetter WL, Rajaram R, Antonoff MB, Fujimoto J, Solis LM, Parra ER, Haymaker C, Wistuba II, Swisher SG, Vaporciyan AA, Lin HY, Wang J, Gibbons DL, Jack Lee J, Ajami NJ, Wargo JA, Allison JP, Sharma P, Kadara H, Heymach JV, Sepesi B. Neoadjuvant chemotherapy plus nivolumab with or without ipilimumab in operable non-small cell lung cancer: the phase 2 platform NEOSTAR trial. Nat Med. 2023 Mar;29(3):593-604. doi: 10.1038/s41591-022-02189-0. Epub 2023 Mar 16. PMID 36928818
- [Derived] Cascone T, Weissferdt A, Godoy MCB, William WN Jr, Leung CH, Lin HY, Basu S, Yadav SS, Pataer A, Mitchell KG, Khan MAW, Shi Y, Haymaker C, Solis LM, Parra ER, Kadara H, Wistuba II, Sharma P, Allison JP, Ajami NJ, Wargo JA, Jenq RR, Gibbons DL, Lee JJ, Swisher SG, Vaporciyan AA, Heymach JV, Sepesi B. Nodal immune flare mimics nodal disease progression following neoadjuvant immune checkpoint inhibitors in non-small cell lung cancer. Nat Commun. 2021 Aug 19;12(1):5045. doi: 10.1038/s41467-021-25188-0. PMID 34413300
- [Derived] Cascone T, William WN Jr, Weissferdt A, Leung CH, Lin HY, Pataer A, Godoy MCB, Carter BW, Federico L, Reuben A, Khan MAW, Dejima H, Francisco-Cruz A, Parra ER, Solis LM, Fujimoto J, Tran HT, Kalhor N, Fossella FV, Mott FE, Tsao AS, Blumenschein G Jr, Le X, Zhang J, Skoulidis F, Kurie JM, Altan M, Lu C, Glisson BS, Byers LA, Elamin YY, Mehran RJ, Rice DC, Walsh GL, Hofstetter WL, Roth JA, Antonoff MB, Kadara H, Haymaker C, Bernatchez C, Ajami NJ, Jenq RR, Sharma P, Allison JP, Futreal A, Wargo JA, Wistuba II, Swisher SG, Lee JJ, Gibbons DL, Vaporciyan AA, Heymach JV, Sepesi B. Neoadjuvant nivolumab or nivolumab plus ipilimumab in operable non-small cell lung cancer: the phase 2 randomized NEOSTAR trial. Nat Med. 2021 Mar;27(3):504-514. doi: 10.1038/s41591-020-01224-2. Epub 2021 Feb 18. PMID 33603241
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2, multi-arm study at the University of Texas MD Anderson Cancer Center recruited patients with resectable stage I-IIIA non-small cell lung cancer. It started on 2017-6-9. The first patient gave consent on 2017-6-16. Patients were randomized to either Arm A - Nivolumab or Arm B - Nivolumab + Ipilimumab. After completion, patients were enrolled in Arm C - Nivolumab + Chemotherapy from 2018-12-14 to 2019-7-22 and Arm D - Nivolumab + Ipilimumab + Chemotherapy from 2019-12-30 to 2020-12-1.
Pre-assignment Details: Fifty-three patients were enrolled in Arm A and Arm B, 9 of them were screen failures. Twenty-three patients were enrolled in Arm C, 1 of them was screen failure. Twenty-five patients were enrolled in Arm D, 3 of them were screen failures.
Groups:
- Arm A - Nivolumab: Induction nivolumab 3 mg/kg intravenous on days 1, 15, and 29 followed by surgery within 3 to 6 weeks.
- Arm B - Nivolumab + Ipilimumab: Induction nivolumab 3 mg/kg intravenous (IV) on days 1, 15, and 29 plus ipilimumab 1 mg/kg IV on day 1 followed by surgery within 3 to 6 weeks.
- Arm C - Nivolumab + Chemotherapy: Induction nivolumab 3 mg/kg intravenous (IV) plus cisplatin and docetaxel (or pemetrexed) IV on days 1, 22, and 43 followed by surgery within 3 to 6 weeks.
- Arm D - Nivolumab + Ipilimumab + Chemotherapy: Induction nivolumab 3 mg/kg intravenous (IV) plus cisplatin (or carboplatin) and docetaxel (or pemetrexed) IV on days 1, 22, and 43 plus ipilimumab 1 mg/kg IV on day 1 followed by surgery within 3 to 6 weeks.
Period: Overall Study
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Started | 23 | 21 | 22 | 22
Completed | 21 | 16 | 22 | 20
Not Completed | 2 | 5 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — High surgical risk | 1 | 1 | 0 | 0
Not completed — Progression | 1 | 1 | 0 | 0
Not completed — Lack of resectability | 0 | 1 | 0 | 0
Not completed — Declined surgery | 0 | 1 | 0 | 0
Not completed — No longer surgical candidate | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population. Patients were enrolled in the study after giving consent. Age at enrollment was reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy | Total
Number analyzed (Participants) | 23 | 21 | 22 | 22 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 10 | 13 | 42
  >=65 years | 12 | 13 | 12 | 9 | 46
Age, Continuous [Median (Full Range); unit: YEARS] | 65.9 [46.5 to 83.6] | 66.2 [43.6 to 76.9] | 69.5 [45.6 to 79.3] | 63.1 [39.4 to 77.5] | 65.9 [39.4 to 83.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 12 | 7 | 35
  Male | 15 | 13 | 10 | 15 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 3 | 7
  White | 21 | 16 | 19 | 18 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 22 | 22 | 88
Smoking status [Count of Participants; unit: Participants] — The smoking status of patients at the time of enrollment
  Participants
    Never smoker | 5 | 3 | 5 | 5 | 18
    Former smoker | 14 | 12 | 17 | 13 | 56
    Current smoker | 4 | 6 | 0 | 4 | 14
Stage [Count of Participants; unit: Participants] — The stage of baseline tissue sample from the biopsy of the primary tumor was evaluated according to the TNM classification of the AJCC 7th edition prior to treatment initiation. Patients with higher stage had worse outcome than patients with lower stage. Stage IA was the lowest stage and Stage IIIA was the highest stage in this study.
  Participants
    Stage IA | 4 | 4 | 0 | 0 | 8
    Stage IB | 7 | 8 | 1 | 0 | 16
    Stage IIA | 2 | 5 | 6 | 2 | 15
    Stage IIB | 5 | 0 | 4 | 7 | 16
    Stage IIIA | 5 | 4 | 11 | 13 | 33
Histology [Count of Participants; unit: Participants] — The histology of baseline tissue sample from the primary tumor
  Participants
    Adenocarcinoma | 13 | 13 | 16 | 13 | 55
    Adenosquamous carcinoma | 0 | 1 | 0 | 0 | 1
    Carcinoma with neuroendocrine features | 0 | 0 | 1 | 0 | 1
    Large cell carcinoma | 0 | 0 | 0 | 1 | 1
    Not otherwise specified NSCLC | 0 | 0 | 0 | 2 | 2
    Sarcomatoid carcinoma | 0 | 0 | 0 | 1 | 1
    Squamous cell carcinoma | 10 | 7 | 5 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Major Pathologic Response (mPR)
Description: The percentage of viable tumor cells was averaged across all reviewed tumor slides from the lung resection specimen. The specimen was reviewed by two pathologists and average score was used. Tumors with ≤ 10% of viable tumor cells were considered to have undergone MPR. Patients who did not have surgery was considered to be no MPR.
Time Frame: The lung resection specimen was collected at surgery.
Population: Intention-to-treat popluation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  MPR | 5 | 8 | 7 | 11
  No MPR | 18 | 13 | 15 | 11

2. Secondary Outcome: Pathologic Complete Response (pCR)
Description: The percentage of viable tumor cells was averaged across all reviewed tumor slides from the lung resection specimen. The specimen was reviewed by two pathologists and average score was used. Tumors with 0% of viable tumor cells were considered to have undergone pCR. Patients who did not have surgery was considered to be no pCR.
Time Frame: The lung resection specimen was collected at surgery.
Population: Intention-to-treat popluation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  pCR | 2 | 6 | 4 | 4
  No pCR | 21 | 15 | 18 | 18

3. Secondary Outcome: Radiographic Response
Description: Radiographic response to induction treatment was assessed by RECIST version 1.1
Time Frame: Reassessment after induction therapy
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  CR | 0 | 1 | 0 | 0
  PR | 5 | 3 | 9 | 6
  SD | 15 | 13 | 13 | 14
  PD | 3 | 3 | 0 | 1
  Not evaluable | 0 | 1 | 0 | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization (in Arm A and Arm B) or treatment initiation (in Arm C and Arm D) to the time of death from all causes or to the time of last follow-up.
Time Frame: In Arms A and B, the cutoff date was 2020-2-25. The median follow-up time frame was 22.2 months. In Arms C and D, the cutoff date was 2022-7-18. The median follow-up time frames were 39.2 and 24.0 months respectively
Population: Intention-to-treat population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Months | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached

5. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from randomization (in Arm A and Arm B) or treatment initiation (in Arm C and Arm D) to any progression of primary lung cancer precluding planned surgery, any progression or recurrence (as assessed by imaging and/or histopathologically) of primary lung cancer after surgery, any progression of primary lung cancer in patients without surgery or death from all causes or to the time of last imaging.
Time Frame: as for outcome 4
Population: Intention-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Months | NA [NA to NA] — Not reached | NA [20.1 to NA] — Not reached | NA [21.7 to NA] — Not reached | NA [NA to NA] — Not reached

6. Secondary Outcome: Residual Tumor Classification
Description: The residual tumor (R) classification measures how well the lung tumor was removed by surgery in the anatomic extent. R0 means a complete resection. R1 means a macroscopically complete resection but with microscopic tumor at the surgical margin. R2 means a resection that leaves gross tumor behind. R0 resection is a better surgical outcome than R1, R2 resections and R2 is the worst surgical outcome. The number of R0, R1 and R2 resections were reported among the patients who underwent surgery.
Time Frame: At surgery
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  R0 | 21 | 16 | 20 | 19
  R1 | 0 | 0 | 1 | 1
  R2 | 0 | 0 | 1 | 0
  No surgery | 2 | 5 | 0 | 2

7. Secondary Outcome: 30-day Postoperative Complication
Description: The number of patients who had complications including pulmonary, cardiac, gastrointestinal, genitourinary, neurological, and wound within 30 days after surgery
Time Frame: Within 30 days after surgery
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Complication | 8 | 5 | 7 | 13
  No complication | 13 | 11 | 15 | 7
  No surgery | 2 | 5 | 0 | 2

8. Secondary Outcome: 90-day Mortality
Description: The number of patients who died within 90 days after surgery
Time Frame: Within 90 days after surgery
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Dead | 1 | 0 | 0 | 0
  Alive | 20 | 16 | 22 | 20
  No surgery | 2 | 5 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant from the first study intervention to approximately up to 8 weeks after surgery. After the end of treatment evaluation, all-cause mortality monitoring was performed as permitted by study protocol. In Arms A and B, the cutoff date was 2020-2-25. The median follow-up time frame was 22.2 months. In Arms C and D, the cutoff date was 2022-7-18. The median follow-up time frames were 39.2 and 24.0 months respectively.
Description: The start date, stop date, grade determined by CTCAE version 4, attribution (unrelated, unlikely, possible, probable, definite) to induction treatment of the adverse event were documented
Arm/Group | Arm A - Nivolumab | Arm B - Nivolumab + Ipilimumab | Arm C - Nivolumab + Chemotherapy | Arm D - Nivolumab + Ipilimumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/21 | 3/22 | 3/22
Serious Adverse Events (participants affected / at risk) | 4/23 | 3/21 | 7/22 | 3/22
Other Adverse Events (participants affected / at risk) | 22/23 | 21/21 | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Nivolumab (N=23) | Arm B - Nivolumab + Ipilimumab (N=21) | Arm C - Nivolumab + Chemotherapy (N=22) | Arm D - Nivolumab + Ipilimumab + Chemotherapy (N=22)
Diarrhea/Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (pulmonary embolism) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical Guillain-Barré syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory failutre (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Nivolumab (N=23) | Arm B - Nivolumab + Ipilimumab (N=21) | Arm C - Nivolumab + Chemotherapy (N=22) | Arm D - Nivolumab + Ipilimumab + Chemotherapy (N=22)
ANC increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 4 (4) | 12 (12) | 11 (11)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 7 (7) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Appetite change (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apical pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Atrial arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Auditory hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BUN increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 1 (1) | 12 (12) | 8 (8)
Decreased kidney function (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 11 (11) | 9 (9)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 8 (8) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
EGFRNAA decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Edema right wrist (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0
Endocrine disorders (Type 1 diabetes) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 16 (16) | 8 (8)
Fever (General disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Free T4 decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hair growth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand and foot syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 6 (6) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 6 (6) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LDH increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left Arm weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphatic colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth sore (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (7) | 18 (18) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Node left jaw (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Nose bleed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral thrush (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain left jaw (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain, neuropathic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 9 (9)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (6) | 13 (13) | 6 (6) | 0 (0)
Rash head (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus pressure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disturbance (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Stiffness (Neck shoulders) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrush (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight gain (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT03158129/Prot_SAP_000.pdf